CLINICAL TRIAL: NCT07283133
Title: Effects of Task Specific Circuit Training on Gross Motor Function, Balance, and Quality of Life in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/13
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP); Quality of Life (QOL)
Keywords: Balance; Gross motor function; task-specific circuit training; hemiplegic cp
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-specific circuit training (TSCT) (Experimental): Task-specific circuit training (TSCT) is a high-intensity, progressive programme aimed at improving functional movement through real-life tasks. It consists of 14 workstations, each performing for 1.5 minutes, with a 3-minute rest after completing the full circuit (total ~21 minutes). Activities include standing and reaching, sit-to-stand, stepping, heel/toe raises, squats, stair climbing, balance exercises, core strengthening, and cycling. This structured circuit enhances gross motor skills, balance, coordination, and overall functional performance.
  Interventions: Procedure: Task-Specific Circuit Training (TSCT)
- Conventional physical therapy (Other): Conventional physical therapy for both groups will include stretching exercises, strengthening exercises, and positioning techniques.
  Each spastic muscle will be stretched to the point of mild discomfort, held for 20 seconds, and repeated five times.
  Every child with CP will be assessed individually to identify spastic muscle groups. Each weak muscle will be trained to contract against resistance, with 10 repetitions performed in each session.
  Parents will be advised to make their child sit with legs open on a bench or block, ensuring the heels touch the ground. They will also be instructed to have their child stand against a wall with the legs in moderate abduction and external rotation for 15 minutes daily after exercises.
  Interventions: Procedure: Conventional Physical Therapy

INTERVENTIONS:
Procedure: Task-Specific Circuit Training (TSCT) — Task-specific circuit training program consisting of 14 workstations designed to improve gross motor skills, balance, strength, and functional mobility. Each station includes a specific functional task-such as reaching, sit-to-stand, stepping in different directions, heel-to-toe raises, squatting, straight-leg raises, stair climbing, backward walking, balance-beam walking, core exercises, bridges, opposite-arm/leg raises, side-bridge exercises, and stationary cycling. Progression at each station is achieved by increasing difficulty through adjustments such as varying distances or heights, increasing repetitions, adding weights, altering surfaces (firm/soft), increasing movement speed, reducing squat depth, carrying objects during tasks, or increasing resistance (for cycling). Overall, the program gradually challenges the child's balance, strength, coordination, and motor control by systematically modifying task demands.
  Arms: Task-specific circuit training (TSCT)
Procedure: Conventional Physical Therapy — Conventional physical therapy will include stretching, strengthening, and positioning exercises. Spastic muscles will be stretched to mild discomfort, held for 20 seconds, and repeated five times. Weak muscles will be strengthened with 10 resisted contractions per session. Parents will be advised to seat the child with legs apart on a bench/block with heels supported and to practice wall-standing with legs moderately abducted and externally rotated for 15 minutes daily after exercises.
  Arms: Conventional physical therapy

SUMMARY:
This study investigates how Task-Specific Circuit Training (TSCT) affects gross motor function, balance, and quality of life in children with Cerebral Palsy. Two groups will be compared: one receiving TSCT and the other receiving conventional physiotherapy. Outcome measures, such as the GMFM, Pediatric Balance Scale, and CP-QoL questionnaire, will be recorded before and after a 8-week intervention (40-50 minutes, 3 sessions per week). Participants will be screened using GMFCS levels I-III. The study aims to determine whether TSCT provides greater improvements in functional mobility, postural control, and overall well-being compared to standard therapy.

DETAILED DESCRIPTION:
This study evaluates the effects of a task-specific circuit training program on functional performance in individuals with cerebral palsy. The intervention is based on motor learning principles and emphasizes repetitive, goal-directed, and functionally relevant activities to enhance neuromuscular control and postural stability.

The task-specific circuit training protocol consists of a series of functional workstations targeting gross motor activities commonly required in daily life, including transitional movements, ambulation-related tasks, and static and dynamic balance activities. Exercises are individualized and progressively modified by adjusting task complexity, repetitions, and external support based on participant performance and tolerance. All training sessions are supervised by trained physiotherapists to ensure standardized implementation and safety.

The intervention is delivered over a structured training period with multiple sessions per week. Each session follows a standardized format consisting of a warm-up phase, circuit-based task-specific exercises, and a cool-down phase. The training approach prioritizes active participation, task repetition, and functional relevance to promote motor performance and functional independence.

The study examines changes in functional outcomes following the intervention period to determine the clinical utility of task-specific circuit training as a rehabilitation strategy for individuals with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Spastic Hemiplegic Cerebral Palsy.
* Age range 5-12 years.
* GMFCS Levels I-III, indicating the ability to walk independently or with assistance.
* Modified Ashworth Scale score 0 to ≤ 2.
* Sufficient cognitive ability to participate in training and follow instructions.

Exclusion Criteria:

* Modified Ashworth Scale (MAS) score greater than 2 in key muscle groups.
* GMFCS Levels IV-V, indicating inability to walk.
* History of frequent seizures.
* Inability to follow verbal or visual instructions, or presence of severe cognitive impairment.
* Recent orthopedic surgery or Botulinum Toxin (Botox) injections.
* Severe musculoskeletal abnormalities such as spinal deformities, hip dislocation, or significant contractures limiting movement.
* Any respiratory, metabolic, or cardiovascular condition that may limit safe participation.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2025-09-13 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Gross motor function | 8 week
  Gross motor function is measured by GMFM-88. These are the gold-standard tools for evaluating changes in gross motor abilities in CP children. It helps to evaluate changes in motor skills over time or after intervention.
  Assesses gross motor functions such as lying, rolling, sitting, crawling, standing, walking, running, and jumping. 80-100% Near-normal motor function / mild CP 40-80% Moderate motor impairment < 40% Severe motor impairment
Balance | 8 week
  Balance is measured by the Pediatric Balance Scale (PBS). Contains 14 tasks such as standing, reaching, turning, and transferring. Scores range from 0 to 5. 50-56 Normal or near-normal balance 33-49 Moderate balance impairment 0-32 Poor balance / high fall risk
Cerebral Palsy Quality of Life | 8 week
  Quality of life is measured by CP QOL (Cerebral Palsy Quality of Life Questionnaire). It measures domains such as: Social well-being, Emotional well-being, Participation, Pain and disability, Access to services, Family health. Scores range 0-100 > 70 High QOL 50-70 Moderate QOL < 50 Low QOL

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan